CLINICAL TRIAL: NCT04474808
Title: Investigation of the Effectiveness of a Foot Cream Containing L-arginine Compared to a Foot Cream Containing Urea for the Care of Dry and Cracked Skin
Brief Title: Foot Cream for the Care of Dry and Cracked Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Bionatural GmbH (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, Director, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Foot cream trial
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine-containing foot cream (Experimental): The participants apply one foot (randomized assignment) with the L-arginine-containing foot cream twice a day (morning and evening) over a period of six weeks.
  Interventions: Other: L-Arginin containing foot cream
- Urea-containing foot cream (Active Comparator): The participants apply one foot (randomized assignment) with the Urea-containing foot cream twice a day (morning and evening) over a period of six weeks.
  Interventions: Other: Urea-containing foot cream

INTERVENTIONS:
Other: L-Arginin containing foot cream — The participants apply one foot (randomized assignment) with the study cream twice a day (morning and evening) over a period of six weeks.
  Arms: L-arginine-containing foot cream
Other: Urea-containing foot cream — The participants apply one foot (randomized assignment) with the control cream twice a day (morning and evening) over a period of six weeks.
  Arms: Urea-containing foot cream

SUMMARY:
In healthy people, but especially in people with diabetes, dry and cracked skin areas on the feet can occur. It is believed that the appearance of dry skin results from a deterioration in the barrier function due to (neuro-) physiological or neuropathic changes in the skin. The standard treatment for skin dryness mainly consists of appropriate care with moisturizing cleaning and care products to protect and restore the barrier function of the skin. Care products containing urea are often used here because urea reduces the feeling of dry and cracked skin due to its moisturizing, keratoplastic, bacteriostatic, antifungal, itch-relieving and proteolytic properties. However, urea-containing preparations can cause painful skin irritation and burning pain on cracked, injured or extremely inflamed skin. Comparable care effects with better tolerance were postulated for care creams enriched with L-arginine. Therefore, a newly developed cream containing 4% L-arginine for the care of dry and cracked skin should be tested in comparison to a conventional care cream containing 5% urea.

DETAILED DESCRIPTION:
Since the participants are recruited during a routine visit to the outpatient clinic or the study center of the West German Diabetes and Health Center (WDGZ), no visits to the study center are necessary as part of the study.

recruitment

* Check the inclusion and exclusion criteria
* Clarification with written confirmation
* Demographic data (including contact details)
* Completing the foot care questionnaire (week 0)
* Delivery of the two creams for the next six weeks
* Handover questionnaires for week 2, 4 and 6 including prepaid envelopes

Study phase (6 weeks) Participants cream their feet with the study creams twice a day (morning and evening) over a period of six weeks. Since there is no contact with medical study staff during this time, undesirable study effects on the behavior of the participants remain minimal.

The use of other creams or care products (except for cleaning) on the feet is not permitted during the study phase.

Questionnaires Foot care questionnaires are completed after two, four, and six weeks and sent to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Appearance of dry and cracked skin on the feet
* Spoken and written knowledge of German
* A written declaration of consent is available

Exclusion Criteria:

* Severe psychiatric illness (e.g. dementia, schizophrenia), which affects the understanding of what the clinical trial is about and the willingness to adhere to the prescribed study procedure
* The appearance of dry skin or itching as a result of an acute or chronic illness (other than diabetes mellitus) or as a side effect of taking medication
* Treatment with systemically or locally acting drugs, in which side effects of skin changes or changes in the barrier function of the skin occur and can thus influence the study results
* Acute clinical symptoms of skin disease on the feet or legs
* Lower limb amputation or acute diabetic foot syndrome
* deep wounds on the feet or legs (Wagner stage 2 to 5)
* Lack of mobility to be able to carry out daily skin care
* Known allergy or intolerance to individual ingredients of the foot care products used in the study
* Restricted legal capacity or legal support
* Participation in other clinical trials with - approved or non-approved - drugs or medical devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Feet Care Feelings | 6 weeks
  Change in the foot care score (according to the questionnaire) after 6 weeks to feel to what extent the skin is dry, rough, scaly, cracked, irritated or reddened, itchy, painful, smooth, tender, soft or horny.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West German Centre of Diabetes and Health
Locations (1):
- West German Centre of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No